CLINICAL TRIAL: NCT00943215
Title: The Proposed Study Entails a Follow-up of All the Completers for 2 Years With Visits Timed 3, 6, 12 and 24 Months After Completion of the 2-year CALERIE II Intervention.
Brief Title: How Participants Behave and Respond on Their Own After Completing a 2-year Intervention of Calorie Restriction
Acronym: CALERIE2-FU
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Eric Ravussin, Princiapal Investigator, Pennington Biomedical Research Center
Other Study IDs: PBRC 29012; NIH U01 AG20478 (Other: NIA)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Excessive Diet Restriction
Keywords: CALERIE II Follow-up

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to gain knowledge about how participants behave and respond on their own after completing a 2-year intervention of calorie restriction.

DETAILED DESCRIPTION:
You will not be assigned to any particular group during the Follow-Up Study. In the Follow-Up study there is no diet intervention. You will not be asked to follow a calorie-restricted diet or any other diet.

Month 3 and Month 6 (Outpatient Visits)following procedures performed:

* Blood pressure, heart rate, temperature, Weight & Waist Measurement
* Medication and medical history
* Blood draw (approximately ½ cup)
* DEXA and QuickScan
* Psychological assessment questionnaires reviewed for completeness
* Body Acceptability Morph Test (BAM)
* Review of 7-day food diary

Month 12 and Month 24 (Outpatient Visits) procedures performed:

* Collection of 4 urine samples
* Dosing with doubly labeled water (DLW)
* DEXA and QuickScan
* Eat breakfast and lunch
* Receive 7-day food diary
* Psychological assessment questionnaires
* Body Acceptability Morph Test (BAM)

Fourteen days after Month 12 and Month 24 (Overnight Inpatient Visits) following procedures performed:

* Collection of 2 urine samples
* Blood pressure, heart rate, temperature, Weight & Waist Measurement
* Blood draw (approximately ½ cup)
* Medication and medical history
* Review of 7-day food diary
* Metabolic Chamber
* Resting Metabolic Rate (RMR)

ELIGIBILITY:
Inclusion Criteria:

* You may qualify to participate in this study only if you completed the CALERIE II study at Pennington Biomedical Research Center.

Exclusion Criteria:

* If you were not a participant in CALERIE II at Pennington Biomedical Research Center, you are ineligible.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants that completeded the CALERIE II study at Pennington Biomedical Research Center.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Calorie Restriction | 2-year
  The purpose of this study is to gain knowledge about how participants behave and respond on their own after completing a 2-year intervention of calorie restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Ravussin, PhD, Principal Investigator — Pennington Biomedical Research Center

REFERENCES:
- [Derived] Marlatt KL, Redman LM, Burton JH, Martin CK, Ravussin E. Persistence of weight loss and acquired behaviors 2 y after stopping a 2-y calorie restriction intervention. Am J Clin Nutr. 2017 Apr;105(4):928-935. doi: 10.3945/ajcn.116.146837. Epub 2017 Mar 8. PMID 28275127
- [Derived] Lam YY, Redman LM, Smith SR, Bray GA, Greenway FL, Johannsen D, Ravussin E. Determinants of sedentary 24-h energy expenditure: equations for energy prescription and adjustment in a respiratory chamber. Am J Clin Nutr. 2014 Apr;99(4):834-42. doi: 10.3945/ajcn.113.079566. Epub 2014 Feb 5. PMID 24500151